CLINICAL TRIAL: NCT05288179
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Phase III Clinical Trial of Efficacy and Safety of Pirfenidone Capsules in the Treatment of Pneumoconiosis
Brief Title: Efficacy and Safety of Pirfenidone Capsules in the Treatment of Pneumoconiosis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Continent Pharmaceutical Co, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GNI-F647-202101
Record Dates: First submitted 2022-02-17; First posted 2022-03-21 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Pneumoconiosis
MeSH Terms: conditions — Pneumoconiosis | interventions — pirfenidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pirfenidone group (Experimental): Patient takes pirfenidone 3 times a day，Week 1, 2 capsules/time; Week 2, 4 capsules/time; Week 3-52, 6 capsules/time
  Interventions: Drug: Pirfenidone Capsules
- placebo group (Placebo Comparator): Patients take a placebo 3 times a day，Week 1, 2 capsules/time; Week 2, 4 capsules/time; Week 3-52, 6 capsules/time
  Interventions: Drug: placebo capsules

INTERVENTIONS:
Drug: Pirfenidone Capsules — After randomization, the experimental group took pirfenidone capsules 3 times a day，Week 1, 2 capsules/time; Week 2, 4 capsules/time; Week 3-52, 6 capsules/time
  Other Names: F647
  Arms: Pirfenidone group
Drug: placebo capsules — After randomization, the experimental group took placebo capsules 3 times a day，Week 1, 2 capsules/time; Week 2, 4 capsules/time; Week 3-52, 6 capsules/time
  Other Names: N
  Arms: placebo group

SUMMARY:
This study is a randomized, double-blind, placebo-controlled, multicenter clinical study.

The main purpose of this study was to confirm the efficacy and safety of pirfenidone capsules in the treatment of pneumoconiosis.

DETAILED DESCRIPTION:
272 patients with pneumoconiosis participated in the 52-week study and were randomized to pirfenidone or placebo.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 18~70 years old (including 18 years old and 70 years old), gender is not limited.

  2. Diagnosed with silicosis or coal worker's pneumoconiosis, in line with GBZ 70-2015 "Diagnosis of Occupational Pneumoconiosis".

  3. Forced vital capacity at screening percentage of predicted value %FVC≥40% and <80% 4. The percentage of carbon monoxide dispersion in the predicted value at the time of screening %DLCO≥30% and <80%.

  5.HRCT at screening showed diffuse interstitial changes in the lungs. 6. Patients voluntarily participated in this trial, with good compliance, and had the ability to understand and sign informed consent before the study.

Exclusion Criteria:

* 1. Those who do not meet any of the inclusion criteria. 2. Those who have received lung lavage therapy within 3 months and plan to receive lung lavage therapy during the trial.

  3. ALT or AST > 3 times ULN. 4. TBiL > 2 times ULN. 5. Creatinine clearance <30 mL/min. 6. Patients with co-infection or high fever within 4 weeks prior to screening, including but not limited to acute bronchitis, pneumonia, sinusitis, urinary tract infection, or cellulitis.

  7. Combined with tuberculosis or lung cancer. 8. Significant pulmonary arterial hypertension requiring parenteral therapy with epoprostenol/treprostinil or severe right heart failure determined by the investigator to be unsuitable to participate in the trial.

  9. Severe cardiovascular disease with one of the following conditions:
  1. Severe hypertension within 6 weeks and uncontrolled with treatment (≥160/100 mmHg);
  2. Myocardial infarction within 6 months;
  3. Unstable angina within 6 months. 10. Coagulation parameters: International normalized ratio (INR) > 2, prothrombin time (PT) prolongation > 1.5 times ULN.

     11. Other conditions or comorbidities that may interfere with testing procedures (eg, intolerance to interruption of supplemental oxygen during pulmonary function tests) or, based on the investigator's judgment, that may interfere with trial participation or that may put patients at risk.

     12. Patients with dysphagia or clinical signs of malabsorption or who require parenteral nutrition.

     13. With active peptic ulcer. 14. History of thrombotic events (including stroke and transient ischemic attack) within 12 months.

     15. Use of cytotoxic drugs, immunosuppressive drugs, cytokine-modulating drugs, or receptor antagonist drugs such as azathioprine, cyclophosphamide, cyclosporine, etanercept, infliximab, white Triene antagonists, methotrexate, tacrolimus, TNF-α inhibitors and tyrosine kinase inhibitors TKIs and other drugs.

     16. Use of interferon, bisbenzylisoquinoline alkaloids (tetrandrine), polyethylene pyrimidine nitroxide (gramsilpine), quinape phosphate, hydroxyquinoline phosphate, aluminum citrate within 1 month before randomization , nintedanib, or high-dose acetylcysteine.

     17. Patients who have previously used drugs that may cause pulmonary fibrosis, such as amiodarone, or have been exposed to asbestos, beryllium and other substances, or exposed to radioactive environments.

     18. Hypersensitivity to the investigational drug or its components (eg, lactose).

     19. Investigator judges that life expectancy due to other medical conditions is < 2.5 years.

     20. Major surgery planned during treatment. 21. Women who were pregnant, breastfeeding, or planning to become pregnant during the trial.

     22. Women of childbearing age who are unwilling or unable to use a highly effective method of contraception during the 28 days before or 3 months after dosing.

     23. According to the researcher, the patient is either alcohol or drug abuser. 24. mentally ill. 25. Those who participated in clinical trials of other drugs within 3 months. 26. Investigators judged to be unfit to participate in the trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Estimated)
Dates: Start 2022-06-07 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Changes in pulmonary function FVC% | 52 weeks
  Change in FVC % (FVC % predicted) at 52 weeks of treatment

SECONDARY OUTCOMES:
Pulmonary function FVC | 52 weeks
  Changes in FVC (L) at 52 weeks of treatment
Changes in lung function DLco% | 52 weeks
  Change in DLco% at 52 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Huaping Dai, Dr, Principal Investigator — China-Japan Friendship Hospital
Locations (1):
- Beijing China-Japan Friendship Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No